CLINICAL TRIAL: NCT04978740
Title: Ocular and Palpebral Manifestations of Mastocytosis (MOOMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MOOMA
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Mast Cell Activation Disease; Mast Cell Activation Syndrome; Mast Cell Disease; Urticaria Pigmentosa
MeSH Terms: conditions — Mast Cell Activation Disorders; Mast Cell Activation Syndrome; Urticaria Pigmentosa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants affected by cutaneous and systemic mastocytosis (Experimental): Participants affected by cutaneous and systemic mastocytosis with or without eye disabilities
  Interventions: Other: Ophthalmological examination

INTERVENTIONS:
Other: Ophthalmological examination — Eye examination :
  Ocular tonometry to determine intraocular pressure Refraction assessment Retina examination Slit lamp examination Visual acuity Schirmer's test Corneal topography Funduscopic examination Optical coherence tomography

SUMMARY:
Mastocytosis is a rare condition characterized by an accumulation of mast cell cells in one or more organs such as the liver, bone marrow, spleen and intestines. Its prevalence in the general population is 1 in 10,000.

This pathology is due to the proliferation of a mast cell clone and the excessive release of inflammatory mediators which lead to abnormal tissue infiltration.

To date, there are only a few cases reporting ocular and orbital manifestations of mastocytosis.

Our prospective, interventional and single-center study consist in describing the ocular functional manifestations and ocular surface abnormalities of patients with systemic and cutaneous mastocytosis.

DETAILED DESCRIPTION:
Patient with systemic or cutaneous mastocytosis will be included in the study. Data about organ involvement of mastocytosis will be collected. Participants will be screened with a medical and eye disease history. They will also have an eye exam.

Participants will provide a tears sample.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of mastocytosis
* Male or female, 18 years of age and over
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Disorders that do not allow good visualization of the posterior pole (cataract, intravitreal hemorrhage)
* Patients with another ocular pathology that may bias the results (corneal dystrophy, dysthyroid orbitopathy, retinal pathologies)
* History of refractive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects with mastocytosis presenting eye abnormalities | up to 2 hours
  Number of patients with functional complaints or abnormalities of the surface, orbit, anterior and posterior segment of the eyeball.

SECONDARY OUTCOMES:
Nature and Frequency of eye abnormalities | up to 2 hours
  Details of functional complaints, abnormalities of various specialized examinations such as ocular tonometry to determine intraocular pressure, Refraction assessment, Retina examination, Slit lamp examination, Visual acuity, Schirmer's test, Corneal topography, Funduscopic examination, Optical coherence tomography
Risk factor of eye abnormalities | up to 2 hours
  Significative association with a mastocytosis subtype or certain organ involvements or biological abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Masson Regnault, Poitiers, Nouvelle-Aquitaine, France